CLINICAL TRIAL: NCT06915688
Title: Comparison of Clinical Cure Rate of Doxycycline and Levofloxacin in the Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: A Study Comparing Doxycycline and Levofloxacin for Treating COPD Exacerbations
Acronym: DOLE-COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amina Aslam (Other Government)
Responsible Party: Sponsor-Investigator, Amina Aslam, AAslam, Lahore General Hospital
Organization: Lahore General Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LGH-COPD-2025
Record Dates: First submitted 2025-03-19; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Doxycycline; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): Doxycycline will be given to this group
  Interventions: Drug: Doxycycline
- Arm 2 (Active Comparator): Levofloxacin in copd patients
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Doxycycline — Doxycycline will be given to COPD group 1
  Arms: Arm 1
Drug: Levofloxacin — Levofloxacin given to copd patients
  Arms: Arm 2

SUMMARY:
This study will include patients with chronic obstructive pulmonary disease (COPD) who present with an acute exacerbation. Participants will be randomly assigned to receive either doxycycline or levofloxacin for 5 days. The aim is to compare how effective each antibiotic is in improving symptoms after 2 days of treatment.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate the effectiveness of two antibiotics-doxycycline (a tetracycline) and levofloxacin (a fluoroquinolone)-in the treatment of acute exacerbations of chronic obstructive pulmonary disease. Participants will be assigned to one of the two treatment groups and will receive either doxycycline 100 mg twice daily or levofloxacin 500 mg once daily for 5 days. The primary outcome is clinical cure. This will be evaluated 2 days after completion of antibiotic therapy, based on symptom resolution and laboratory markers.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed cases of COPD Exacerbation of COPD Able to provide Written consent No anti biotic taken with in past 4 weeks

Exclusion Criteria:

* hypersensitivity to any drugs Pneumonia evidence on xray/ hrct chest Any other pulmonary condition e.g asthma Pregnancy/breast feeding Taking treatment for other active infections

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Cure Rate | 7 days
  1. A decrease in the respiratory rate by 20% from the baseline measurement.
  2. Restoration of Oxygen saturation levels to within the range of 88-92% on room air.
  3. CRP<10ng/ml
  4. decrease in sputum quantity
  5. reduction in body temperature below 99•F
  6. TLC <11,000

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided